CLINICAL TRIAL: NCT04992351
Title: Wide-awake Local Anesthesia and no Tourniquet (WALANT) in Plastic Surgery: Indications, Clinical Applications and Outcomes
Brief Title: Wide-awake Local Anesthesia and no Tourniquet (WALANT) in Plastic Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Ioannina (Other)
Responsible Party: Principal Investigator, Konstantinos Seretis, Ass. Professor of Plastic Surgery, University Hospital, Ioannina
Other Study IDs: 11335
Record Dates: First submitted 2021-07-13; First posted 2021-08-05 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Upper Limb Wound; Lower Limb Wound; Anesthesia, Local
Keywords: WALANT; plastic surgery; upper limb; lower limb

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WALANT group: WALANT was used exclusively as anesthesia method for the operation
  Interventions: Procedure: WALANT
- control: tourniquet with regional or general anesthesia was used for the operation
  Interventions: Procedure: WALANT

INTERVENTIONS:
Procedure: WALANT — WALANT as anesthesia method for upper and lower limb palstic surgery operations

SUMMARY:
Wide-awake local anesthesia no tourniquet (WALANT) was proposed and performed in hand operations.

Aim of this study is to present the use of WALANT in operations performed on the upper and lower limbs, evaluate its efficacy in terms of feasibility, total operation time, total operating room time, bleeding, patient discomfort and satisfaction and control for potential drawbacks. The hypothesis is that WALANT is a viable option in common operations performed by plastic surgeons on the upper and lower limbs.

DETAILED DESCRIPTION:
Wide-awake local anesthesia no tourniquet (WALANT) was proposed and performed in hand operations. Little has been studied, regarding its indications and efficacy in general plastic surgery operations.

Aim of this study is to present the use of WALANT in operations performed on the upper and lower limbs, evaluate its efficacy in terms of feasibility, total operation time, total operating room time, bleeding, patient discomfort and satisfaction and control for potential drawbacks. The hypothesis is that WALANT is a viable option in common operations performed by plastic surgeons on the upper and lower limbs.

A prospective study will be conducted comparing the use of WALANT in operations performed on the upper and lower limbs to the traditional use of tourniquet with general or regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* upper or lower limb operation
* indication for flap or skin grafting
* operated by the principal investigator

Exclusion Criteria:

* other concomitant operations performed
* known allergy to any of the ingredients of local anesthesia mixture

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who undergo general plastic surgery operations in the upper or lower limb
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
total operation time | through operation completion
  the difference between skin incision and skin closure in minutes
operation theatre time | through operation completion with exit from the operation theatre
  the difference between entry and exit of the patient from the operation theatre in minutes
Patient satisfaction | at 8 weeks
  estimated by a 10-point visual analogue scale (1-10, 10 is the best outcome)
feasibility of the WALANT method | through operation completion
  percentage of cases, which could not be completed under WALANT with conversion to the traditional method of anesthesia

SECONDARY OUTCOMES:
complications | at 8 weeks
  number and type of complications in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Plastic Surgery Department, Ioannina, Greece

IPD SHARING:
Plan to Share IPD: No